CLINICAL TRIAL: NCT05993780
Title: An Evaluation of End-Expiratory Lung Volume and Pulmonary Mechanics With Different PEEP Levels in Mechanical Ventilation in ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Selvinaz Yüksel Tanrıverdi, Specialist, Department of Anesthesiology and Reanimation, MD, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PamukkaleUSyuksel-001
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Ards
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARDS patient (Other): 14 patients with ARDS were included in the study. It was planned as a single group.
  Interventions: Other: No drugs or biologial agents were used in our trial

INTERVENTIONS:
Other: No drugs or biologial agents were used in our trial — Before the measurement, a recruitment maneuver was performed for 30-40 s at a PEEP level of 20 cmH2O. At four different PEEP levels of 15, 10, 5, and 0 cmH2O, a decreasing PEEP trial was performed, and the measurement results were recorded.The measurement time at each PEEP level was chosen as 10 minutes. At the end of the measurement, static compliance was measured by applying an end-inspiratory pause. Respiratory system elastance,static strain volume gain was calculated.The estimated lung volume recovered was calculated using the formula ∆EELV - (∆PEEP x Compliance PEEPlow) and compared with the volume gain.

SUMMARY:
ARDS management is quite complex, and mortality is high. PEEP titration is very important in mechanical ventilation. However, the most appropriate approach for PEEP titration has yet to be determined. Currently, the emphasis is on focused PEEP implementation. The present study aimed to evaluate the volume gain at different PEEP levels over the pressure-volume curve, the changes in EELV measured by the modified multiple nitrogen wash-out/wash-in technique, and the compliance with respiratory mechanics.

14 adult ARDS patients undergoing invasive mechanical ventilation were included in the study. According to the Berlin Criteria, There were two mild, seven moderates, and five severe ARDS patients. FRC and EELV with decreased PEEP titration estimates (5 cmH2O) were measured by the multiple nitrogen wash-out/washin technique. Gain and compliance values were measured over the dynamic pressure-volume curves created by the intracheal pressure sensor.

DETAILED DESCRIPTION:
The present study was conducted in the Anesthesiology and Reanimation Intensive Care Units of Pamukkale University Hospital with the approval of Pamukkale University Non-Interventional Clinical Research Ethics Committee dated 13.07.2021 and 13th board meeting numbered 60116787-020/83538. Between August 2021 and August 2022, 17 patients were included over 18 years of age who met the Berlin criteria and were diagnosed with ARDS sedated, intubated, and mechanically ventilated. Informed written consent was obtained from the relatives.

Patients included in the study were connected to a CARESCAPE R860 (GE Healthcare) mechanical ventilator. Rocuronium bromide was administered intravenously to eliminate the spontaneous respiratory effort and opioids for sedation. Tidal volume was adjusted as 6 ml/kg according to the estimated body weight; the respiratory rate was adjusted to ensure normocarbia in blood gas analysis; FiO2 was adjusted as PaO2 55 to 80 mmHg; end-inspiratory pause was adjusted to 20%, and inspiratory/expiratory ratio was adjusted as 1:2.

The ECOV-X (GE Healthcare) module was attached to the ventilator for gas measurements and allowed to warm up. A spirometer kit was inserted between the Y-piece in the ventilator circuit and the bacterial/viral filter with heat and moisture-retaining properties. An intratracheal pressure sensor was inserted to measure pressure levels independent of circuit and tube resistance and to evaluate them on the SpiroDynamics (GE Healthcare) application. EELV was measured with the ECOV-X (GE Healthcare) module using a modified NMBW technique with the change in FiO2. EELV was calculated using VO2 (oxygen consumption) and VCO2 (carbon dioxide production). After all the connections were completed, the VO2 and VCO2 values of the patients were measured. The PEEP titration procedure called Lung INview (GE Healthcare) was initiated in patients whose values stabilized within 30 min. Before the measurement, a recruitment maneuver was performed for 30-40 s at a PEEP level of 20 cmH2O. At four different PEEP levels of 15, 10, 5, and 0 cmH2O, a decreasing PEEP trial was performed, and the measurement results were recorded.

For the same PEEP levels, the shunt fraction decreases when a decreasing PEEP maneuver is used instead of an increasing PEEP maneuver. This suggests that the relationship between optimal PEEP and maximum compliance may be more accurate. Therefore, decreasing PEEP trials was preferred as the study protocol.

The measurement time at each PEEP level was chosen as 10 minutes. At the end of the measurement, static compliance was measured by applying an end-inspiratory pause. Tidal volume, peak, and driving pressure were recorded at each step. Respiratory system elastance was calculated using the equation by Henderson et al.(respiratory system elastance = driving pressure/tidal volume). The static strain was calculated using the equation using the tidal volume at the relevant PEEP value (static strain =VPEEP/FRC). The pressure-volume curve generated by the intratracheal pressure sensor at each PEEP level was evaluated using the SpiroDynamics application. A dynamic compliance curve was generated during the analysis, and volume changes in this curve were determined at each PEEP level. The difference in EELV at two different PEEP levels during a descending PEEP trial was calculated as ∆EELV, and the difference between ∆EELV and the volume derived from the pressure-volume curve was calculated as "volume gain" (gain = ∆EELV - volume derived from the curve). The estimated lung volume recovered was calculated using the formula ∆EELV - (∆PEEP x Compliance PEEPlow) and compared with the volume gain. The efficiency of the volume gains concept as an indicator of the volume gained by alveolar recruitment and its role in personalized PEEP titration was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ARDS according to the Berlin criteria
* Berlin definition criteria: (1) presence of acute hypoxemic respiratory failure, (2) onset within 7 days of insult, or or new (within 7 days) or worsening respiratory symptoms; (3) bilateral opacities on chest x-ray or CT not fully explained by effusions, lobar or lung collapse, or nodules; and (4) cardiac failure not primary cause of acute respiratory failure.

Exclusion Criteria:

* Patients with severe cardiovascular instability (Mean arterial pressure <60 mmHg , Pulse <45 or >150), Patients with pneumothorax, Patients who have undergone pneumonectomy operation, Patients with Lung Transplantation, Patients with thoracic deformity, ARDS patients with cor pulmonale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Does volume gain indicate recruited lung volume? | Patients were ventilated for 10 minutes at each PEEP level.Measurement was taken after 10 minutes.]
  A dynamic compliance curve was generated during the analysis, and volume changes in this curve were determined at each PEEP level. The difference in EELV at two different PEEP levels during a descending PEEP trial was calculated as ∆EELV, and the difference between ∆EELV and the volume derived from the pressure-volume curve was calculated as "volume gain" (gain = ∆EELV - volume derived from the curve). The estimated lung volume recovered was calculated using the formula ∆EELV - (∆PEEP x Compliance PEEPlow) and compared with the volume gain.

SECONDARY OUTCOMES:
Static compliance correlation with volume gain. | Patients were ventilated for 10 minutes at each PEEP level.Measurement was taken after 10 minutes.
  After measuring the volume gain, its correlation with static compliance was examined. The measurement time at each PEEP level was chosen as 10 minutes. At the end of the measurement, static compliance was measured by applying an end-inspiratory pause
Calculation of respiratory system elastance and its correlation with volume gain. | Patients were ventilated for 10 minutes at each PEEP level.Measurement was taken after 10 minutes.
  Respiratory system elastance was calculated using the equation (respiratory system elastance = driving pressure/tidal volume).
Examination of the relationship between static strain and volume gain. | Patients were ventilated for 10 minutes at each PEEP level.Measurement was taken after 10 minutes.
  Static strain; calculated by the ratio of tidal volume to FRC at the relevant PEEP level.
Investigation of the correlation between driving pressure and volume gain | Patients were ventilated for 10 minutes at each PEEP level.Measurement was taken after 10 minutes.
  During the measurements, volume gain and driving pressure at different PEEP levels were recorded and their correlations were examined.

OTHER OUTCOMES:
Hemodynamic parameters of patient with ARDS were measured during different PEEP measurement. | Measurements were taken after 10 minutes of ventilating at the PEEP level.
  Systolic blood pressure, diastolic blood pressure and heart rate, peripheral oxygen saturation at different PEEP levels were recorded.
Arterial blood gas analysis | Measurements were taken after 10 minutes of ventilating at the PEEP level.
  At all PEEP levels, pH, PaO2 (mmHg), PaCO2 (mmHg), SaO2 (%) were measured in arterial blood gas.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No